CLINICAL TRIAL: NCT01347749
Title: Mindfulness and Self-Compassion Meditation for Combat Posttraumatic Stress Disorder: Randomized Controlled Trial and Mechanistic Study
Brief Title: Mindfulness and Present Centered Therapies for PTSD: Efficacy and Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: VA Ann Arbor Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Anthony King, Research Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-08-2-0208
Record Dates: First submitted 2011-04-27; First posted 2011-05-04 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Meditation; Mindfulness; Compassion; Group Psychotherapy; Emotional Regulation; fMRI
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Emotional Regulation | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness & Compassion Meditation-based Exposure Therapy (Experimental): A 16 week group psychotherapy intervention involving PTSD psychoeducation, breathing exercises and relaxation, and Mindfulness and Self-compassion meditation exercises in session and daily at home, and Mindfulness-based in vivo exposure exercises.
  Interventions: Behavioral: Mindfulness & Compassion Meditation-based Exposure Therapy
- Present Centered Therapy for PTSD (Active Comparator): This is a more standard from of group psychotherapy (talk therapy) which focusses on current symptoms and stressors
  Interventions: Behavioral: Present Centered Therapy for PTSD

INTERVENTIONS:
Behavioral: Mindfulness & Compassion Meditation-based Exposure Therapy — A 16 week group psychotherapy intervention involving PTSD psychoeducation, breathing exercises and relaxation, and Mindfulness and Self-compassion meditation exercises in session and daily at home, and Mindfulness-based in vivo exposure exercises.
  Other Names: Mindfulness-based Exposure therapy
  Arms: Mindfulness & Compassion Meditation-based Exposure Therapy
Behavioral: Present Centered Therapy for PTSD — This 16 week, active group psychotherapy involves PTSD psychoeducation, supportive listening, and focusses on current stressors and PTSD symptoms.
  Other Names: Present Centered Group Therapy
  Arms: Present Centered Therapy for PTSD

SUMMARY:
This project will study whether a new therapy that includes the practice of forms of meditation is helpful for combat veterans returning from deployments in Iraq or Afghanistan suffering with posttraumatic stress disorder (PTSD). "Mindfulness meditation" cultivates present-focused, non-judgmental attention to ones body, emotions, and thoughts, and is proposed to lead to a greater sense of well-being and acceptance and better tolerance of painful and distressing emotions. "Compassion" and "loving-kindness" meditations help stabilize positive emotions like love and compassion, and may also be helpful for chronic pain, and possibly depression and PTSD.

This study will compare a 16 week psychotherapy group for PTSD involving Mindfulness and Self-compassion meditation, with a more standard form of group psychotherapy known as "Present-centered group therapy". Both therapies will be conducted at the VA Ann Arbor PTSD clinic by VA psychotherapists. (The study is also approved by the IRB of the VA Ann Arbor). Combat veterans will be randomly assigned to either the Meditation or the standard group psychotherapy. All patients will also receive fMRI brain scans before and after the therapy, as well as assessment interviews before, at 8 weeks, and immediately post-therapy, and at 3 mo and 6 mo follow-ups. Saliva cortisol and measures of attention will also be obtained at each assessment.

DETAILED DESCRIPTION:
Background: "Mindfulness meditation" is an ancient "Mind-Body" attentional technique for cultivating present-focused, non-judgmental attention to sensory, interoceptive, emotional, and cognitive processes. It is proposed to lead to a greater sense of well-being and acceptance, greater cognitive flexibility, and better tolerance of painful and distressing physical, emotional, and cognitive phenomena. Our group has found a model of emotional meta-awareness leads to decreased amygdala and increased medial prefrontal cortex (mPFC) activation. Mindfulness meditation has also been suggested to work by volitionally altering self-related cognitive/emotional processing to shift away from the predominate 'narrative' (and potentially ruminative) mode to a more 'experiential', present-centered mode in which arising sensations, percepts, emotions, and cognitions can be perceived with greater equanimity and flexibility. Mindfulness-based Stress Reduction (MBSR) is helpful for coping with chronic pain, fibromyalgia, and distress and anxiety associated with major medical disorders, and Mindfulness-based Cognitive Therapy (MBCT) for preventing depression relapse in patients. "Compassion meditation" is likewise an ancient practice for cultivating and stabilizing a sense of pro-social, empathic, kind/loving and compassionate regard to one's self and others, and in the Tibetan tradition, is based upon a 'foundation' of mindfulness. A single small trial found a loving-kindness meditation improved chronic lower back pain symptoms, and neuroimaging studies have found effects on emotional neurocircuitry.

Objective/Hypothesis: We hypothesize that practice of mindfulness and Tibetan self-compassion meditation by PTSD patients will lead to 1.) improvement in PTSD and other symptoms and quality of life 2.) improved emotional regulation, attentional control, increased 'mindfulness' and self-compassion, and 3.) strengthening of mPFC circuits during emotional provocation. There are theoretical considerations and limited empirical data that mindfulness and Tibetan compassion meditation may be useful for combat-related PTSD, which is marked by exaggerated emotional responses and distress to trauma memories and cues, distressing guilt and self-blame, and emotional dysregulation; however, the acceptability and efficacy of mindfulness and Tibetan compassion meditation not been demonstrated in combat PTSD. A pilot study at the Ann Arbor VA PTSD Clinic adapted a psychotherapy using mindfulness meditation, mindful stretching exercises, and Tibetan compassion meditation for use in combat PTSD, and found significant reductions in 'avoidant' PTSD symptoms and self-blame cognitions compared to a treatment-as-usual group. Importantly, we were also able to identify some obstacles to acceptability that have provided our group with greater insight and experience into how to acceptably and effectively deliver meditation programs to combat veterans seeking treatment for PTSD. PTSD neuroimaging studies implicate deficits during emotional provocation in medial prefrontal cortex (mPFC), associated with emotional regulation.

Specific Aims:

Aim 1. Further develop a manualized group psychotherapy based on mindfulness and Tibetan self-compassion meditation for combat PTSD.

Aim 2. Formally test our meditation intervention for PTSD in a randomized controlled trial.

Aim 3. Utilizing a 'translational design', perform a pilot study of fMRI neuroimaging to determine the effects of meditation on neurocircuitry underlying emotional regulation that may mediate therapeutic effects

Study Design: We will develop a manual for our meditation incorporating input from qualitative data from patients and an expert advisory board including meditation and PTSD therapy experts. We will adapt a present-centered therapy group as a control intervention, controlling for hours of therapist contact. We will randomly assign PTSD patients to either meditation or present-cetnered therapy, with pre- post, 3 mo, and 6 mo follow-up assessments with validated measures of PTSD and psychiatric symptoms, quality of life, "mindfulness", emotional regulation, and trauma-related maladaptive cognitions. We will also perform a pilot study of fMRI neuroimaging to determine the effects of meditation on neurocircuitry underlying emotional regulation that may mediate therapeutic effects. Validated emotional and social cognition neuroimaging paradigms will be used to examine specific effects of mindfulness meditation on mPFC and cortico-limbic neurocircuitry.

Impact: This research will examine the efficacy of a highly novel treatment approach for PTSD, and also specific neural mechanisms of emotional regulation and how they may be altered by effortful rehearsal of alternate emotion regulation and emotion induction techniques. It may thus lead to improved treatment and understanding of therapeutic mechanisms involving emotional regulation.

ELIGIBILITY:
Inclusion Criteria:

* Combat veteran serving in Iraq or Afghanistan Has PTSD (CAPS score > 40)

Exclusion Criteria:

* Suicidality Substance dependence not in treatment Personality disorder taking medications that interfere with stress hormone measures

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2011-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale | pre-therapy, and post-therapy (week 16)
  is an interview measure of PTSD severity and the primary outcome measure for the study. Current PTSD will be assessed in relation to the OEF/OIF war-zone trauma that is currently most upsetting. The CAPS has excellent psychometrics. Completion requires about 45 minutes.

SECONDARY OUTCOMES:
PTSD Checklist (PCL-C) | pre-therapy, and post-therapy (week 16)
  is a 17-item self-report assessment of PTSD severity using a 5-point scale, from 1 (not at all) to 5 (very often). It has good reliability and validity.
Posttraumatic Cognitions Inventory (PTCI) | pre-therapy, and post-therapy (week 16)
  PTCI is a 36-item assessment of negative thoughts about the self, negative thoughts about the world, and self-blame. It has good psychometrics and has been related to change in PTSD symptoms with treatment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan